CLINICAL TRIAL: NCT04510220
Title: Open-label, Observational, Prospective, 9-month Study to Assess the Efficacy of Ofatumumab on Microglia in Patients With Relapsing Forms of Multiple Sclerosis
Brief Title: 9-month Study to Assess the Efficacy of Ofatumumab on Microglia in Patients With Relapsing Forms of Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, TARUN SINGHAL, Associate Professor of Neurology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P002078
Record Dates: First submitted 2020-07-31; First posted 2020-08-12 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — ofatumumab; N-fluoroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects diagnosed with relapsing forms of multiple sclerosis (Experimental): We plan to enroll 10 subjects with relapsing MS. All enrolled subjects will receive Ofatumumab 20 mg every 4 weeks, subcutaneously for 9 months during the study. Loading doses will be administered initially at 1, 7 and 14 days. During the study period, all enrolled subjects will undergo five PET scans using [F-18] PBR06 at day 0, 5, 28, 90 (3 Months) and 273 (9 Months) after starting treatment with Ofatumumab.
  Interventions: Drug: Ofatumumab; Drug: [F-18]PBR06

INTERVENTIONS:
Drug: Ofatumumab — Ofatumumab (OMB157) is a fully human anti-CD20 monoclonal antibody (mAb) self-administered by a once-monthly subcutaneous injection that is in development for MS. Ofatumumab drug product (also referred as OMB157) is formulated as 20 mg/0.4 mL (50 mg/mL) solution for injection, provided in autoinjectors, for subcutaneous administration. The autoinjectors contain a small overfill to allow for a complete withdrawal of the labeled amount (20 mg) of ofatumumab.
  Other Names: OMB157
Drug: [F-18]PBR06 — PET radiopharmaceutical. Subjects will undergo [F-18]PBR06-PET (microglial activation).
  Other Names: [18F]PBR06

SUMMARY:
We aim to assess the effect of Ofatumumab on microglial activation using [F-18]PBR06 PET in MS patients in relation to changes in serum markers, MRI abnormalities and clinical impairment longitudinally over 9 months.

Specific Aims:

Specific Aim 1: To determine the effect of Ofatumumab on microglial activation in MS over 9 months.

Specific Aim 2: To determine the time course of effect of Ofatumumab on microglial activation and its relationship with peripheral B-cell depletion, serum neurofilament light (sNfL) chain and glial-fibrillary acid protein (GFAP) levels and other serum biomarkers

Specific Aim 3: To determine the relationship of PET changes following Ofatumumab initiation with 3T MRI changes and clinical parameters.

DETAILED DESCRIPTION:
Design: This is an open-label, observational, prospective, 9-month follow-up study to assess the efficacy of ofatumumab on microglia pathology in patients with MS, as measured by changes in microglial activation in the lesional and non-lesional, normal appearing white matter, cortical and subcortical grey matter, and peri-plaque area of chronic lesions in the brain.

Initial Visit:

During the first visit, subjects will be administered the screening questionnaire (if that has not already been done over telephone). Subjects will review and eventually sign the consent form. They will be administered a physical examination, clinical assessment and standardized questionnaires for cognitive testing and/or other co-morbidities. In addition, blood samples will be drawn for genotype testing, infection screening, complete blood count and liver function test.

Demographics, physical examinations and neurologic assessments will be conducted at Brigham MS Center, Brigham and Women's Hospital, 60 Fenwood Road, Boston, MA 02115.

Genotype Testing:

Blood sample drawn on the initial screening visit will be used to obtain genomic DNA for genotyping for polymorphism within the TSPO gene on chromosome 22q13.2, using a Taqman assay. High affinity and medium affinity binders will be included in the study, whereas low affinity binders will be excluded from the study.

PET Scanning:

For this study, all subjects will undergo five separate visits for [F-18]PBR06 PET scans, one visit before starting Ofatumumab treatment (day 0 baseline) and four more visits at approximately 5, 28, 90 and 273 days after initiating treatment. During the PET scan visits, all women subjects of child bearing age will undergo a stat quantitative serum hCG pregnancy test and only women with a negative test will undergo the radiopharmaceutical injection. The radiotracers will be produced using standardized procedures. At the time of imaging, the subjects will be positioned in the gantry of a high-resolution PET/CT camera. Head alignment will be made, relative to the canthomeatal line, using projected laser lines whose positions are known with respect to the slice positions of the scanner. A head support apparatus will be used to minimize head motion. Dynamic data over 120 minutes for PET quantification will be acquired, according to previously described methods for the tracer.

MRI Scanning:

All subjects will undergo five 3T brain MRIs with and without contrast, one before starting Ofatumumab treatment (day 0 baseline) and four more at 5, 28, 90 and 273 days after initiating treatment. All women will be queried about their pregnancy status, use of contraception and last menstrual period. If a woman is of child bearing potential, she will undergo a urine pregnancy test. Subjects will undergo intravenous gadolinium contrast administration, during all visits. Hence, all women of child bearing potential will undergo urine pregnancy testing for this study.

Clinical Follow-up Visits:

Subjects will come in for five clinical visits, one visit before starting Ofatumumab treatment (day 0 baseline) and four more visits at 5, 28, 90 and 273 days after initiating treatment. However, if the patient meets all inclusion criteria at the screening visit, the screening and baseline visits may occur on the same day. During these visits, subjects will undergo a physical examination, clinical assessment and cognitive assessment. A blood sample will be drawn to determine levels of sNfL, GFAP and other serum biomarkers. Visits will be conducted under the supervision of PI and other board-certified neurologists. Any adverse event reported by the patient or observed by the investigator will be recorded and reviewed at each clinical visit.

Clinical Data:

The following non-imaging, clinical data will be obtained:

Expanded Disability Status Scale (EDSS), Timed 25-feet walk (T25W), 9-Hole Peg Test (9HPT), Four component MS Functional Composite (MSFC-4), Symbol-Digit Modality test (SDMT), cognitive and symptom questionnaires, vision testing, Levels of serum biomarkers.

Clinical Safety Monitoring:

Safety will be assessed at 0, 3, 6, and 9 months of the study including:

* Pregnancy Testing: All women of childbearing potential will undergo a serum pregnancy test at the screening visit and at each of the following scheduled visits to the hospital. The investigator will also review the contraception status of subjects at each visit.
* Electrocardiogram (ECG): An ECG will be performed either at the screening visit or on day 0 clinical visit and at the end of the study.
* Routine labs: Blood samples will be collected at the screening visit and at each visit time point. Blood samples will be assessed for red blood cell count, hemoglobin, hematocrit, platelets, total white blood cell (WBC) count and WBC differential counts (neutrophils, lymphocytes, basophils, eosinophils, monocytes) as well as for electrolytes (Na, K, Cl, bicarbonate, Ca, Mg, P), random glucose, total protein, blood urea nitrogen, albumin, alkaline phosphatase, ALT, AST, GGT, total bilirubin, conjugated bilirubin, creatinine, amylase, C-Reactive protein.
* Samples for total IgM and IgG levels at baseline, 3, 6 and 9 months
* Patient diary review
* Monthly telephone interview

Drug Administration/Dosing:

At the end of the baseline clinic visit, subjects will be instructed by one of the investigators on proper drug administration technique. The first injection of ofatumumab will be performed under the guidance of an appropriately trained healthcare professional in the clinical space at the Brigham MS Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with active, relapsing MS course (defined by Lublin 2014 criteria). Active disease is defined by at least 1 relapse during the previous 1 year or 2 relapses during the previous 2 years or a positive gadolinium-enhancing MRI scan or MRI scan with new or unequivocally enlarging T2 lesions in previous year.
* Age 18 to 60 years
* EDSS 0 to 5.5
* Subjects either untreated or treated with disease modifying therapies other than those listed in exclusion criteria
* Agree to start treatment with ofatumumab and comply with study procedures for the duration of the study
* No other systemic disease or neurological disorders requiring chronic or acute steroid or other immunosuppressive treatment
* No known hypersensitivity reactions to contrast agents
* None of the exclusion criteria

Exclusion Criteria:

* Subjects suspected of not being able or willing to cooperate or comply with study protocol requirements in the opinion of the investigator.
* Subjects with primary progressive MS or SPMS without disease activity.
* Disease duration of more than 10 years in patients with an EDSS score of 2 or less
* Subjects meeting criteria for neuromyelitis optica.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for at least 6 months after stopping study medication. Highly effective contraception methods include:
* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject, if accepted by the local regulation). NOTE: Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal ARE NOT acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking investigational drug. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* For female subjects on the study, the vasectomized male partner should be the sole partner
* Use of oral, (estrogen and progesterone), injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking investigational drug.
* In case local regulations deviate from the contraception methods listed above, local regulations apply and will be described in the ICF.
* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.
* Subjects with active chronic disease (or stable but treated with immune therapy) of the immune system other than MS (e.g. rheumatoid arthritis, scleroderma, Sjögren's syndrome, Crohn's disease, ulcerative colitis, etc.) or with an immunodeficiency syndrome.
* Subjects with a history of the following:

  1. History of any malignancy
  2. History of alcohol or drug abuse
  3. Primary or secondary immunodeficiency
  4. Prior hematopoietic stem cell transplantation
  5. History of transplantation or anti-rejection therapy
* Subjects with the following laboratory abnormalities:

  1. Abnormal CD19+ B-cell levels at screening (defined as CD19 count <110 cells per microliter)
  2. Leukopenia (defined as white blood cell (WBC) count <4000 WBCs per microliter)
  3. Lymphopenia (defined as lymphocyte count <1000 lymphocytes per microliter)
  4. Hypogammaglobulinemia defined as a level of <500mg/dL will be excluded. All subjects with low serum immunoglobulins should be evaluated by a hematologic expert prior to exclusion in the study.
  5. Any abnormality of liver function tests, including ALT/SGPT, AST/SGOT, Alkaline phosphatase, total or direct bilirubin or GGT
* Subjects with active systemic bacterial, viral or fungal infections, or known to have acquired immunodeficiency syndrome (AIDS).
* Subjects with neurological symptoms consistent with PML or confirmed PML.
* Subjects at risk of developing or having reactivation of syphilis or tuberculosis (eg subjects with known exposure to, or history of syphilis, or active or latent tuberculosis, even if previously treated).
* Subjects with low affinity binders (LAB) for TSPO radioligand
* Subjects with abnormal serum creatinine levels (defined as >1.3mg/dL) or Subjects with estimated glomerular filtration rate (eGFR) <30ml/minute
* Patients with history of significant renal disease (dialysis, kidney transplant, single kidney, renal cancer, renal surgery)
* Patient presenting with cardiac disorders defined by at least one of the following conditions:
* Patient with recent cardiac history (within 6 months) of:

  * Acute coronary syndrome
  * Acute heart failure (class III or IV of the NYHA classification)
* History of significant ventricular arrhythmia (persistent ventricular tachycardia, ventricular fibrillation, resuscitated sudden death)
* Patient with history of cardiac failure class III or IV of the NYHA classification
* Patient with history of severe conduction disorders which are not prevented by permanent pacing (atrio-ventricular block 2 and 3, sinoatrial block)
* Syncope without known etiology within 3 months
* Uncontrolled severe hypertension, according to the judgment of the investigator, or symptomatic hypertension
* Subjects with any contraindications to PET/CT or MRI procedures (e.g. claustrophobia, MRI-incompatible implants or pacemakers, renal failure)
* Subjects with any significant or uncontrolled medical comorbidity
* Subjects with active hepatitis B
* Subjects at risk of hepatitis B reactivation (such as subjects with positive HBsAG or anti-Hepatitis B core antibodies) should be evaluated by a liver disease expert before inclusion, or should be excluded
* Subjects treated with other disease modifying treatments within their respective pre-specified washout periods will be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2022-12-28 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Singhal, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham MS Center, 60 Fenwood Road, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Diagnosed With Relapsing Forms of Multiple Sclerosis: We plan to enroll 10 subjects with relapsing MS. All enrolled subjects will receive Ofatumumab 20 mg every 4 weeks, subcutaneously for 9 months during the study. Loading doses will be administered initially at 1, 7 and 14 days. During the study period, all enrolled subjects will undergo five PET scans using [F-18] PBR06 at day 0, 5, 28, 90 (Month 3) and 273 (Month 9) after starting treatment with Ofatumumab.
Period: Overall Study
Arm/Group | Subjects Diagnosed With Relapsing Forms of Multiple Sclerosis
Started | 10
Completed | 9
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Subjects Diagnosed With Relapsing Forms of Multiple Sclerosis: We plan to enroll 10 subjects with relapsing MS. All enrolled subjects will receive Ofatumumab 20 mg every 4 weeks, subcutaneously for 9 months during the study. Loading doses will be administered initially at 1, 7 and 14 days. During the study period, all enrolled subjects will undergo five PET scans using [F-18] PBR06 at 0, 5, 28, 90 and 273 days after starting treatment with Ofatumumab.
Arm/Group | Subjects Diagnosed With Relapsing Forms of Multiple Sclerosis
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 40.2 [23 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Glial Activity Load on PET
Description: The primary endpoint of the study will be the regional glial activity on PET (GALP) measurements at 3 months and 9 months compared to baseline.
  Individualized z-score maps of brain parenchymal microglial activation were generated using a voxel-by-voxel comparison between each subject's 60-90 minute PET standardized uptake value ratio (SUVR) images (globally normalized) and a control dataset of 9 healthy individuals. GALP scores were calculated as the sum of voxel-by-voxel z-scores >4 in a given region divided by the total number of voxels in that region. A z-score of 0 represents the reference population mean. Higher z-scores indicate worse outcomes. A z-score >4 is considered positive and contributes to the average GALP score.
Time Frame: Baseline, 3 Months, and 9 Months
Population: Due to the unavailability of the PET tracer, PET scans at all time points were completed by the first 5 participants only. The baseline, 3 month, and 9 month results for these 5 participants are presented here.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Subjects Diagnosed With Relapsing Forms of Multiple Sclerosis
Number analyzed (Participants) | 5
Z-score
  Baseline | 0.968 (0.063)
  3 Months | 0.799 (0.103)
  9 Months | 0.759 (0.171)

2. Secondary Outcome: % CD19 Counts
Description: Peripheral % CD19 (B Cells) counts at 5 days and 9 months compared to baseline. This is the proportion of B cells (which express CD19) relative to all lymphocytes.
Time Frame: Baseline, 5 Days, and 9 Months
Population: Due to the unavailability of the PET tracer, PET scans at all time points were completed by the first 5 participants only. The baseline, 5 day, and 9 month results for these 5 participants are presented here.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Subjects Diagnosed With Relapsing Forms of Multiple Sclerosis
Number analyzed (Participants) | 5
Percentage
  Baseline | 14.70 (9.75)
  5 Days | 0.98 (1.10)
  9 Months | 0.04 (0.09)

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up, up to 9 months.
Groups:
- Subjects Diagnosed With Relapsing Forms of Multiple Sclerosis: We plan to enroll 10 subjects with relapsing MS. All enrolled subjects will receive Ofatumumab 20 mg every 4 weeks, subcutaneously for 9 months during the study. Loading doses will be administered initially at 1, 7 and 14 days. During the study period, all enrolled subjects will undergo five PET scans using [F-18] PBR06 at 0, 5, 28, 90 and 273 days after starting treatment with Ofatumumab.
  Ofatumumab (OMB157) is a fully human anti-CD20 monoclonal antibody (mAb) self-administered by a once-monthly subcutaneous injection that is in development for MS. Ofatumumab drug product (also referred as OMB157) is formulated as 20 mg/0.4 mL (50 mg/mL) solution for injection, provided in autoinjectors, for subcutaneous administration. The autoinjectors contain a small overfill to allow for a complete withdrawal of the labeled amount (20 mg) of ofatumumab.
  PET radiopharmaceutical. Subjects will undergo [F-18]PBR06-PET (microglial activation).
Arm/Group | Subjects Diagnosed With Relapsing Forms of Multiple Sclerosis
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Diagnosed With Relapsing Forms of Multiple Sclerosis (N=10)
Scanning related issues (General disorders) | 3 — pain, discomfort, soreness, spasms, minor panic attack
Injection related issues (Product Issues) | 8 — chills, body aches, fever, headache, bruising, numbness, myalgia, itchiness, redness, swelling, fatigue, nausea
IV related issues (General disorders) | 3 — discomfort, bruising

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT04510220/Prot_SAP_000.pdf